CLINICAL TRIAL: NCT02520245
Title: Companion Study for Patients Who Completed Participation in a REGN2810 (Anti-PD-1) Clinical Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1425
Record Dates: First submitted 2015-08-05; First posted 2015-08-11 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-05

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — cemiplimab

ARMS (1):
- Open-Label (Experimental)
  Interventions: Drug: REGN2810

INTERVENTIONS:
Drug: REGN2810 — Patients will receive REGN2810 by intravenous (IV) infusion

SUMMARY:
This study has been designed to collect long-term follow-up information for patients who received REGN2810 in other clinical studies and to allow re-treatment for eligible patients.

ELIGIBILITY:
The target population for this study is patients who have participated in any REGN2810 clinical study.

Inclusion Criteria for Patients Receiving Re-treatment:

1. Tolerated prior treatment with REGN2810 with no unacceptable toxicity (except select reversible irAEs) requiring discontinuation of REGN2810
2. Developed documented progressive disease after first demonstrating clinical benefit from their initial treatment
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
4. ≥18 years old
5. Hepatic function:

   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN; if liver metastases ≤ 3 x ULN)
   * Transaminases ≤ 3 x ULN (or ≤ 5.0 x ULN, if liver metastases)
   * Alkaline phosphatase (ALP) ≤ 2.5 x ULN (or ≤ 5.0 x ULN, if liver metastases)
   * For patients with hepatic metastases or hepatic malignancies, exclude patients with concomitant 3 x ULN ≤ aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 5 x ULN and 1.5 x ULN ≤ total bilirubin ≤ 3 x ULN
6. Renal function: Serum creatinine ≤ 1.5 x ULN
7. Bone marrow function:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Platelet count ≥ 75 x 10^9/L

Inclusion Criteria for Patients who Will not Receive Re-treatment:

Patients must have completed participation in any REGN2810 clinical study.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from receiving re-treatment with REGN2810:

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for irAEs.
2. Patients who experienced an irAE in while participating in another REGN2810 protocol who were unable to have their corticosteroid dose reduced to <10 mg per day prednisone equivalent within 12 weeks of toxicity.
3. Patients who developed ≥ Grade 2 uveitis in a prior REGN2810 protocol
4. Immunosuppressive corticosteroid doses (> 10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of REGN2810
5. Active infection requiring therapy, including known infection with human immunodeficiency virus, or active infection with hepatitis B or hepatitis C virus.
6. History of pneumonitis within the last 5 years.
7. Any investigational or antitumor treatment within 30 days prior to the initial administration of REGN2810.
8. History of documented allergic reactions or acute hypersensitivity reaction attributed of Grade ≥ 3 severity during or directly following an REGN2810 infusion
9. Known allergy to doxycycline or tetracycline. (precaution due to presence of trace components in REGN2810)
10. Breast-feeding
11. Positive serum pregnancy test
12. History within the last 5 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
13. Acute or chronic psychiatric problems that, under the evaluation of the investigator, make the patient ineligible for participation
14. Unwilling to practice adequate contraception during the study until 6 months after the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival, from the first dose of study drug administered in the parent REGN2810 clinical study to death or date of last censoring | up to 8 years
Safety measured by the number of patients with AEs, AEs leading to discontinuation, SAEs, drug-related AEs, Immune-related adverse events (irAEs), and death as outcome. | up to 8 years
  Safety includes the number of patients with AEs, AEs leading to discontinuation, SAEs, drug-related AEs, Immune-related adverse events (irAEs), and death as outcome.

SECONDARY OUTCOMES:
Response duration (time from best overall response of partial or complete response, to time to first documented disease progression) | up to 8 years
Duration of disease control (time from best overall response of SD as well as PR and CR to time to first do documented disease progression) | up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (9):
- United States (9):
  - City of Hope National Medical Center, Duarte, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Laura & Isaac Perlmutter Cancer Center, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - START South Texas Accelerated Research Therapeutics, San Antonio, Texas